CLINICAL TRIAL: NCT01385280
Title: A Pilot Study Of Estradiol Followed By Exemestane For Post-Menopausal Hormone Receptor Positive Metastatic Breast Cancer After Prior Failed Endocrine Therapy: Reversing Endocrine Resistance
Brief Title: Pilot Study Estradiol Followed by Exemestane Hormone Receptor + Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0906-04; NCI-2010-02366 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3P30CA023074 (NIH)
Record Dates: First submitted 2011-06-22; First posted 2011-06-30 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Progesterone Receptor Positive Tumor; Recurrent Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol; exemestane; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral therapeutic estradiol once daily on days 1-3, twice daily on days 4-7, and thrice daily on days 8-90. Beginning on day 98, patients receive oral exemestane once daily in the absence of disease progression or unacceptable toxicity. Also laboratory biomarker analysis and enzyme-linked immunosorbent assay will be taken for correlative studies.
  Interventions: Biological: therapeutic estradiol; Drug: exemestane; Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay

INTERVENTIONS:
Biological: therapeutic estradiol — Given orally (PO)
  Other Names: Aquadiol; Dimenformon; Diogyn; Diogynets; ESDL
Drug: exemestane — Given PO
  Other Names: Aromasin; FCE-24304; PNU 155971
Other: laboratory biomarker analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA

SUMMARY:
RATIONALE: Estrogen can cause the growth of tumor cells. Hormone therapy using therapeutic estradiol may fight breast cancer by lowering the amount of estrogen the body makes. Though estradiol initially produces stimulation of ER+ cancer cells, both laboratory and some clinical experience indicate that it may have the opposite effect on such cells, once they have become resistant to estrogen deprivation. In laboratory models, there is death of the "resistant" population after estradiol treatment, followed by restoration of sensitivity of the remaining cells to estrogen deprivation, as with an aromatase inhibitor. Exemestane may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving therapeutic estradiol together with exemestane may kill more tumor cells.

PURPOSE: This clinical trial studies therapeutic estradiol and exemestane in treating post-menopausal patients with hormone receptor-positive metastatic breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess feasibility and toxicity associated with estradiol followed by exemestane in the treatment of estrogen receptor positive metastatic breast cancer patients failing prior aromatase inhibitor therapy.

II. Exploratory analysis of bio-correlates which will evaluate the mechanism of action of this treatment combination: changes in serum M-30, a marker of mitochondrial apoptosis; changes in number of circulating tumor cells (CTC); changes in CTC expression of ER, IGF1-R, and M-30.

III. Exploratory analysis of Progression Free Survival (PFS).

OUTLINE: Patients receive oral therapeutic estradiol once daily on days 1-3, twice daily on days 4-7, and thrice daily on days 8-90. Beginning on day 98, patients receive oral exemestane once daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with metastatic carcinoma of the breast; post-menopausal, as defined by at least one of the following: at least 12 months without spontaneous menstrual bleeding, history of bilateral salpingo-oophorectomy with or without hysterectomy, age > 55 with hysterectomy with or without oophorectomy, serum Follicle-stimulating hormone (FSH) in post-menopausal range within 4 weeks of registration.
* Positive for estrogen receptor (ER) or progesterone receptor (PgR) with positivity defined as immunohistochemical staining in >= 10% of cells
* Either measurable disease by RECIST or non-measurable evaluable disease; tests to evaluate disease (measurable and non-measurable) must be completed within 28 days prior to registration; these will include a CT scan of the chest/abdomen/pelvis and a bone scan; patients with effusions or ascites as the only sites of disease are ineligible
* Performance status of 0-2 by Zubrod criteria
* Patients must have a baseline CA15-3 or CA 27.29 measurement for future comparison, but any baseline value is acceptable
* Patients must have had prior aromatase inhibitor (AI) therapy in the metastatic setting (any number of prior AI is allowed, this may have been any of the AI's), or have developed metastatic disease on adjuvant AI therapy; prior treatment with tamoxifen and/or fulvestrant is also allowed; patients must not have been previously treated with estradiol for metastatic breast cancer
* Patients must be able to take oral medications
* Patients must be informed of the investigational nature of this study and give written informed consent in accordance with institutional and federal guidelines
* Patients must consent to the serum and CTC blood specimen submissions

Exclusion Criteria:

* Planning to receive concomitant chemotherapy, hormone therapy (including hormone replacement therapy), radiation therapy, or antibody therapy for malignancy while receiving protocol treatment, with the single exception of trastuzumab; concomitant trastuzumab will be allowed for Her-2 positive patients who were previously on trastuzumab; patients who have had previous radiotherapy must complete treatment within 4 weeks of registration, and have recovered from acute toxicity from radiation; patients with prior cytotoxic chemotherapy for metastatic disease will not be eligible
* Known hypersensitivity or intolerance to estradiol, aromatase inhibitors, or aspirin; patients must not have a history of aspirin-induced GI bleeding within the past 3 years
* Known untreated brain or CNS metastases due to the risk of bleeding on aspirin during estradiol
* History of deep vein thrombosis, pulmonary embolism, or other clot requiring anticoagulation; patients must not have a known inherited hypercoagulable disorder
* History of decompensated congestive heart failure, unstable angina, or uncontrolled psychiatric illness which would limit compliance with the protocol treatment
* Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Livingston, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Chalasani P, Stopeck A, Clarke K, Livingston R. A pilot study of estradiol followed by exemestane for reversing endocrine resistance in postmenopausal women with hormone receptor-positive metastatic breast cancer. Oncologist. 2014 Nov;19(11):1127-8. doi: 10.1634/theoncologist.2014-0306. Epub 2014 Sep 26. PMID 25260365

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 4 Toxicity
Description: Such as deep vein thrombosis requiring hospitalization or pulmonary embolism
Time Frame: By day 90
Population: Study was terminated - the PI is deceased. Attempts were made to locate the data but it seems that data were never fully collected/analyzed.
Arm/Group | Arm I
Number analyzed (Participants) | 0

2. Secondary Outcome: Patients With Change in Serum M-30 (a Marker of Mitochondrial Apoptosis) With Treatment
Time Frame: At baseline and on days, 8, 30, 60, and 90
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

3. Secondary Outcome: Patients With Change in Number of Circulating Tumor Cells (CTC) With Treatment
Time Frame: At baseline and on days 8, 90, and 180
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

4. Secondary Outcome: Patients With Change in Circulating Tumor Cells (CTC) Expression of M-30 With Treatment
Time Frame: At baseline and on days 8, 90, and 180
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Circulating Tumor Cells (CTC) ER Expression With Treatment
Time Frame: At baseline and on days 8, 90, and 180
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Circulating Tumor Cells (CTC) IGF1R Expression With Treatment
Time Frame: At baseline and on days 8, 90, and 180
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

7. Secondary Outcome: Median Time From Entry on Study to Progression of Disease
Description: In weeks
Time Frame: Up to 1.5 years
Population: as for outcome 1
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=13)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=13)
Abdominal Pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight Loss (Metabolism and nutrition disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes